CLINICAL TRIAL: NCT06651567
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Flexible-dose Study of the Efficacy, Safety, and Tolerability of ITI-1284 in Patients With Agitation Associated With Alzheimer's Dementia
Brief Title: A Study to Assess the Efficacy and Safety of ITI-1284 in the Treatment of Agitation Associated With Alzheimer's Dementia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITI-1284-101
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Agitation Associated With Alzheimer's Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ITI-1284 (Experimental): ITI-1284 10 mg or 20 mg rapidly disintegrating tablet, taken once daily, sublingual administration
  Interventions: Drug: ITI-1284
- Placebo (Placebo Comparator): Placebo rapidly disintegrating tablet, taken once daily, sublingual administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ITI-1284 — ITI-1284 10 mg or 20 mg rapidly disintegrating tablet, taken once daily, sublingual administration
  Arms: ITI-1284
Drug: Placebo — Placebo rapidly disintegrating tablet, taken once daily, sublingual administration
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, flexible-dose study of the efficacy, safety, and tolerability of ITI-1284 in patients with agitation associated with Alzheimer's dementia

DETAILED DESCRIPTION:
The study will be conducted in 3 periods:

* Screening Period (up to 4 weeks) during which patient eligibility will be assessed;
* Double-blind Treatment Period (12 weeks) during which all patients will be randomized in a 1:1 ratio to receive either ITI-1284 or placebo;
* Safety Follow-up Period (30 days) during which all patients will return for a safety follow-up visit approximately 30 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Can understand the nature of the trial and protocol requirements and provide signed informed consent, if in the judgement of the Investigator is deemed competent to provide consent or if patient is deemed not competent to provide informed consent, with the patient's assent (if capable), consent may be provided by an appropriate person (eg, patient's Legally Authorized Representative [LAR]) before the initiation of any study-specific procedures in accordance with local regulations;
* Meets clinical criteria for Alzheimer's disease based on 2011 National Institute of Aging-Alzheimer's Association (NIA-AA) dementia criteria and biomarker criteria and either:

  * Has a high likelihood for amyloid pathology consistent with Alzheimer's disease, as confirmed by blood-based biomarker at Screening; or
  * Has historical documentation of cerebrospinal fluid (CSF) biomarker or amyloid positron emission tomography (PET) brain scan;
* Meets all criteria for agitation according to the International Psychogeriatric Association (IPA) consensus definition
* Has clinically meaningful agitation defined as a Neuropsychiatric Inventory-Agitation/Aggression (NPI-AA) domain total score of ≥ 4 at both Screening and Baseline;
* CGI-S score ≥ 4 at Screening and Baseline;
* Has Mini-Mental State Examination, 2nd Edition™: Standard Version (MMSE-2®:SV) score of 6 to 24 at Screening;

Exclusion Criteria:

* Agitation symptoms are attributable to concomitant medications, adverse environmental conditions, substance abuse, or active medical or psychiatric conditions as per Investigator's judgment;
* Has been diagnosed with one or more of the following psychiatric conditions:

  * Schizophrenia, schizoaffective disorder, or other psychotic disorder that is not related to Alzheimer's dementia;
  * Bipolar disorder;
  * Major depressive disorder, unless it is considered stable and treated for at least 8 weeks prior to Screening;
* Has a significant risk for suicidal behavior during the course of their participation in the study, or is considered to be an imminent danger to themselves or others, in the opinion of the investigator, and/or as assessed by Columbia Suicide Severity Rating Scale (C-SSRS); or the patient has had 1 or more suicide attempts within the 2 years prior to Screening;
* The patient has known hypersensitivity or intolerance to ITI-1284 or lumateperone, or to any of their excipients.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Cohen-Mansfield Agitation Inventory (CMAI) total score | Week 12
  The CMAI is a reliable and validated, 29-item caregiver-rating questionnaire to assess agitated behavior in elderly patients. Each item is rated on a 7-point scale of frequency, from "never" (1) to "several times an hour" (7), with 1 being the "best" rating and 7 being the "worst" rating. The minimum possible CMAI total score is 29, and the maximum possible CMAI total score is 203.

SECONDARY OUTCOMES:
Clinical Global Impression-Severity (CGI-S) Score | Week 12
  The CGI-S is a clinician-rated scale to assess a patient's overall mental health. The scale ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients)

CONTACTS AND LOCATIONS:
Locations (55):
- United States (24):
  - Clinical Site, Anaheim, California
  - Clinical Site, Costa Mesa, California
  - Clinical Site, Garden Grove, California
  - Clinical Site, Boca Raton, Florida
  - Clinical Site, Bonita Springs, Florida
  - Clinical Site, Brandon, Florida
  - Clinical Site, Delray Beach, Florida
  - Clinical Site, Doral, Florida
  - Clinical Site, Hialeah, Florida
  - Clinical Site, Homestead, Florida
  - Clinical Site_2, Maitland, Florida
  - Clinical Site, Maitland, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site_2, Miami, Florida
  - Clinical Site_3, Miami, Florida
  - Clinical Site, Orlando, Florida
  - Clinical Site_2, Tampa, Florida
  - Clinical Site, Tampa, Florida
  - Clinical Site, West Palm Beach, Florida
  - Clinical Site, Boston, Massachusetts
  - Clinical Site, Las Vegas, Nevada
  - Clinical Site, Toms River, New Jersey
  - Clinical Site, Raleigh, North Carolina
  - Clinical Site, San Antonio, Texas
- Bulgaria (4):
  - Clinical Site, Lovech
  - Clinical Site, Pleven
  - Clinical Site, Sofia
  - Clinical Site, Stara Zagora
- Croatia (3):
  - Clinical Site_2, Zagreb
  - Clinical Site_3, Zagreb
  - Clinical Site, Zagreb
- Czechia (5):
  - Clinical Site, Brno
  - Clinical Site, Choceň
  - Clinical Site, Kutná Hora
  - Clinical Site, Pilsen
  - Clinical Site, Prague
- Romania (3):
  - Clinical Site, Bucharest
  - Clinical Site, Sânpetru
  - Clinical Site, Sibiu
- Serbia (5):
  - Clinical Site_2, Belgrade
  - Clinical Site, Belgrade
  - Clinical Site, Kovin
  - Clinical Site, Niš
  - Clinical Site, Novi Kneževac
- Slovakia (6):
  - Clinical Site, Banská Bystrica
  - Clinical Site, Bratislava
  - Clinical Site, Košice
  - Clinical Site, Krompachy
  - Clinical Site, Svidník
  - Clinical Site, Vranov nad Topľou
- Spain (5):
  - Clinical Site, Albacete
  - Clinical Site, Barcelona
  - Clinical Site, Málaga
  - Clinical Site, Zamora
  - Clinical Site, Zaragoza

IPD SHARING:
Plan to Share IPD: No